CLINICAL TRIAL: NCT06524284
Title: Feasibility of Self-treatment of Painful Diabetic Neuropathy Using Electrical Vasomotor Nerve Stimulation
Acronym: HOME-EVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurecon BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOME-EVNS-01
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-04

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- EVNS treatment (Experimental): EVNS, see intervention
  Interventions: Device: Releaf

INTERVENTIONS:
Device: Releaf — 10 days/35 minutes per day EVNS (non-invasive electrostimulation) treatment on lower legs and feet by the subject or its caregiver after instruction by the podiatrist.

SUMMARY:
Electrical stimulation with EVNS (Electrical Vasomotor Neuro Stimulation), a methodology used by a specific group of neurostimulators known under various names, has proven its benefit in Painful Diabetic Neuropathy (PDN). However, due to the impaired mobility from Diabetic Neuropathy, a part of subjects did not finish the 10 days treatment in the outpatient clinic. Another part of the target group decided not to participate at all for the same reason.

The current study investigates the feasibility, safety and performance of a newly developed EVNS device, called Releaf™, optimised for HOME treatment,

ELIGIBILITY:
Inclusion Criteria:

* Painful Diabetic Neuropathy (DN4 positive) and insufficiently treated with any combination of 2 of the following drugs: Duloxetine (Cymbalta), venlafaxine (Efexor), ami- or nortriptyline, gabapentine, pregabaline (Lyrica) or the use of carbamazepine or capsaïcine (Qutenza).
* Both feet are present
* Able and willing to complete the treatments in 10 days in a row and completion of questionnaires.
* Being in a mental and physical state to perform home self-treatment with Releaf™ for 10 consecutive days, if necessary with adequate assistance of caregiver.
* Being in a mental and physical state to understand and complete the informed consent form as well as the research questionnaires.

Exclusion Criteria:

* In case of other evident causes for painful neuropathy,
* Currently participating in another interventional investigational study
* Significant peripheral arterial disease,
* Active foot ulceration or other skin conditions that prevent the application of electrodes on the skin
* Current alcohol or other substance abuse (use of alcohol over the recommended limits of less than 21 units of alcohol per week in men and 14 units in women, Trimbos Intitute),
* Epilepsy,
* Pregnancy,
* Presence of a medical device based on electrical stimulation, cardiac pacemaker and/or implantable cardioverter defibrillator or any other active implant
* Allergy to electrode contact area or to the adhesive substance of the electrode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Side-effects | Day 1-10
  The number and severity of reported side-effects of HOME-EVNS, gathered via telephonic consulting on treatment day 1,3 and 8 and via user-initiated incoming calls to the PI
Successful treatment cycles | Day 11
  The successful treatment cycles applied at home, defined as cycles with at least 8/10 successful (full 35 minutes) treatment sessions, derived from the adherence determined by recording device usage and intensity setting which is downloaded from device after its retrieval
Reported usability | Day 10
  Usability by the User Questionnaire
Use of helpdesk | Day 1-10
  The number of help requests to service desk.

SECONDARY OUTCOMES:
Neuropathic pain | Before start, after 1 month, after 3 months
  Neuropathic Pain Symptom Inventory (NPSI) filled in by subject
Quality of life score | Before start, after 1 month, after 3 months
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) QoL filled in by subject

CONTACTS AND LOCATIONS:
Overall Officials: Ben Imholz, PhD, MD, Principal Investigator — Neurecon BV
Locations (1):
- Neurecon, Vught, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alleman CJ, Westerhout KY, Hensen M, Chambers C, Stoker M, Long S, van Nooten FE. Humanistic and economic burden of painful diabetic peripheral neuropathy in Europe: A review of the literature. Diabetes Res Clin Pract. 2015 Aug;109(2):215-25. doi: 10.1016/j.diabres.2015.04.031. Epub 2015 May 6. PMID 26008721
- [Background] Azmi S, Petropoulos IN, Ferdousi M, Ponirakis G, Alam U, Malik RA. An update on the diagnosis and treatment of diabetic somatic and autonomic neuropathy. F1000Res. 2019 Feb 15;8:F1000 Faculty Rev-186. doi: 10.12688/f1000research.17118.1. eCollection 2019. PMID 30828432
- [Background] Bevilacqua M, Dominguez LJ, Barrella M, Barbagallo M. Induction of vascular endothelial growth factor release by transcutaneous frequency modulated neural stimulation in diabetic polyneuropathy. J Endocrinol Invest. 2007 Dec;30(11):944-7. doi: 10.1007/BF03349242. PMID 18250616
- [Background] Bocchi L, Evangelisti A, Barrella M, Scatizzi L, Bevilacqua M. Recovery of 0.1Hz microvascular skin blood flow in dysautonomic diabetic (type 2) neuropathy by using Frequency Rhythmic Electrical Modulation System (FREMS). Med Eng Phys. 2010 May;32(4):407-13. doi: 10.1016/j.medengphy.2010.02.004. Epub 2010 Mar 6. PMID 20207576
- [Background] Bosi E, Conti M, Vermigli C, Cazzetta G, Peretti E, Cordoni MC, Galimberti G, Scionti L. Effectiveness of frequency-modulated electromagnetic neural stimulation in the treatment of painful diabetic neuropathy. Diabetologia. 2005 May;48(5):817-23. doi: 10.1007/s00125-005-1734-2. Epub 2005 Apr 15. PMID 15834546
- [Background] Bosi E, Bax G, Scionti L, Spallone V, Tesfaye S, Valensi P, Ziegler D; FREMS European Trial Study Group. Frequency-modulated electromagnetic neural stimulation (FREMS) as a treatment for symptomatic diabetic neuropathy: results from a double-blind, randomised, multicentre, long-term, placebo-controlled clinical trial. Diabetologia. 2013 Mar;56(3):467-75. doi: 10.1007/s00125-012-2795-7. Epub 2012 Dec 13. PMID 23238789
- [Background] Crasto W, Altaf QA, Selvaraj DR, Jack B, Patel V, Nawaz S, Murthy N, Sukumar N, Saravanan P, Tahrani AA. Frequency Rhythmic Electrical Modulation System (FREMS) to alleviate painful diabetic peripheral neuropathy: A pilot, randomised controlled trial (The FREMSTOP study). Diabet Med. 2022 Mar;39(3):e14710. doi: 10.1111/dme.14710. Epub 2021 Nov 3. PMID 34605077
- [Background] D'Souza RS, Barman R, Joseph A, Abd-Elsayed A. Evidence-Based Treatment of Painful Diabetic Neuropathy: a Systematic Review. Curr Pain Headache Rep. 2022 Aug;26(8):583-594. doi: 10.1007/s11916-022-01061-7. Epub 2022 Jun 18. PMID 35716275
- [Background] Dworkin RH, Turk DC, Revicki DA, Harding G, Coyne KS, Peirce-Sandner S, Bhagwat D, Everton D, Burke LB, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA, Melzack R. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009 Jul;144(1-2):35-42. doi: 10.1016/j.pain.2009.02.007. Epub 2009 Apr 7. PMID 19356853
- [Background] Emerson GG, Segal SS. Electrical activation of endothelium evokes vasodilation and hyperpolarization along hamster feed arteries. Am J Physiol Heart Circ Physiol. 2001 Jan;280(1):H160-7. doi: 10.1152/ajpheart.2001.280.1.H160. PMID 11123230
- [Background] Gibson W, Wand BM, Meads C, Catley MJ, O'Connell NE. Transcutaneous electrical nerve stimulation (TENS) for chronic pain - an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2019 Apr 3;4(4):CD011890. doi: 10.1002/14651858.CD011890.pub3. PMID 30941745
- [Background] Gorczyca-Siudak D, Dziemidok P. The 8-Week Efficacy of Frequency Rhythmic Electrical Modulated System (FREMS) as an Add-on Therapy in the Treatment of Symptomatic Diabetic Peripheral Polyneuropathy. Int J Environ Res Public Health. 2022 Dec 22;20(1):111. doi: 10.3390/ijerph20010111. PMID 36612433
- [Background] Gunter C, Delbeke J, Ortiz-Catalan M. Correction to: Safety of long-term electrical peripheral nerve stimulation: review of the state of the art. J Neuroeng Rehabil. 2020 Jun 15;17(1):77. doi: 10.1186/s12984-020-00695-1. PMID 32539841
- [Background] Imholz B, Heijster J, Tahrani A, Kooy A. Treatment of Painful Diabetic Neuropathy Using Frequency Rhythmic Electro Magnetic Neural Stimulation (FREMS); Effectiveness in Daily Practice. Diabetes Metab Syndr Obes. 2023 May 11;16:1383-1391. doi: 10.2147/DMSO.S401727. eCollection 2023. PMID 37197061
- [Background] Johnson MI, Paley CA, Jones G, Mulvey MR, Wittkopf PG. Efficacy and safety of transcutaneous electrical nerve stimulation (TENS) for acute and chronic pain in adults: a systematic review and meta-analysis of 381 studies (the meta-TENS study). BMJ Open. 2022 Feb 10;12(2):e051073. doi: 10.1136/bmjopen-2021-051073. PMID 35144946
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Strand NH, Burkey AR. Neuromodulation in the Treatment of Painful Diabetic Neuropathy: A Review of Evidence for Spinal Cord Stimulation. J Diabetes Sci Technol. 2022 Mar;16(2):332-340. doi: 10.1177/19322968211060075. Epub 2021 Nov 29. PMID 34842478
- [Background] Tesfaye S, Wilhelm S, Lledo A, Schacht A, Tolle T, Bouhassira D, Cruccu G, Skljarevski V, Freynhagen R. Duloxetine and pregabalin: high-dose monotherapy or their combination? The "COMBO-DN study"--a multinational, randomized, double-blind, parallel-group study in patients with diabetic peripheral neuropathic pain. Pain. 2013 Dec;154(12):2616-2625. doi: 10.1016/j.pain.2013.05.043. Epub 2013 May 31. PMID 23732189
- [Background] Wang EJ, Berninger LE, Komargodski O, Smith TJ. Painful Diabetic Neuropathy - Spinal Cord Stimulation, Peripheral Nerve Stimulation, Transcutaneous Electrical Nerve Stimulation, and Scrambler Therapy: A Narrative Review. Pain Physician. 2022 Nov;25(8):E1163-E1173. PMID 36375183
- [Background] Zeng H, Pacheco-Barrios K, Cao Y, Li Y, Zhang J, Yang C, Fregni F. Non-invasive neuromodulation effects on painful diabetic peripheral neuropathy: a systematic review and meta-analysis. Sci Rep. 2020 Nov 5;10(1):19184. doi: 10.1038/s41598-020-75922-9. PMID 33154432
- [Background] Zhao M, Bai H, Wang E, Forrester JV, McCaig CD. Electrical stimulation directly induces pre-angiogenic responses in vascular endothelial cells by signaling through VEGF receptors. J Cell Sci. 2004 Jan 26;117(Pt 3):397-405. doi: 10.1242/jcs.00868. Epub 2003 Dec 16. PMID 14679307
- [Background] Ziegler D, Tesfaye S, Spallone V, Gurieva I, Al Kaabi J, Mankovsky B, Martinka E, Radulian G, Nguyen KT, Stirban AO, Tankova T, Varkonyi T, Freeman R, Kempler P, Boulton AJ. Screening, diagnosis and management of diabetic sensorimotor polyneuropathy in clinical practice: International expert consensus recommendations. Diabetes Res Clin Pract. 2022 Apr;186:109063. doi: 10.1016/j.diabres.2021.109063. Epub 2021 Sep 20. PMID 34547367
- [Background] Zucatti KP, Teixeira PP, Wayerbacher LF, Piccoli GF, Correia PE, Fonseca NKO, Moresco KS, Guerra BA, Madure MG, Farenzena LP, Frankenberg AD, Brietzke E, Halpern B, Franco O, Colpani V, Gerchman F. Long-term Effect of Lifestyle Interventions on the Cardiovascular and All-Cause Mortality of Subjects With Prediabetes and Type 2 Diabetes: A Systematic Review and Meta-analysis. Diabetes Care. 2022 Nov 1;45(11):2787-2795. doi: 10.2337/dc22-0642. PMID 36318674